CLINICAL TRIAL: NCT01846208
Title: Oral Desensitization to Egg With Subsequent Induction of Sustained Unresponsiveness for Egg-Allergic Children Using Baked Egg or Egg Oral Immunotherapy (OIT)
Brief Title: Baked Egg or Egg Oral Immunotherapy for Children With Egg Allergy
Acronym: CoFAR7
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hugh A Sampson, MD (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Consortium of Food Allergy Research (Other)
Responsible Party: Sponsor-Investigator, Hugh A Sampson, MD, Director, Jaffe Food Allergy Institute, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 04-1271; U19AI066738 (NIH); CoFAR7 (Other: Consortium of Food Allergy Research)
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Results first posted 2018-10-30 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Food Allergy
Keywords: Egg Allergy; Egg Oral Immunotherapy; Food Allergy
MeSH Terms: conditions — Food Hypersensitivity; Egg Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Egg OIT Randomized (Experimental): Subjects who passed a baked egg oral food challenge (OFC) at baseline were randomized to receive egg oral immunotherapy (OIT) in the form of egg white solid with up to four oral food challenges as directed by protocol.
  Interventions: Drug: Egg Oral Immunotherapy
- Baked Egg Randomized (Experimental): Subjects who passed a baked egg oral food challenge (OFC) at baseline were randomized to receive baked egg in the form of home-baked goods and "safe" commercial products with up to four oral food challenges as directed by the protocol.
  Interventions: Drug: Baked Egg
- Egg OIT Assigned (Experimental): Subjects who failed a baked egg oral food challenge (OFC) at baseline were assigned to receive egg oral immunotherapy (OIT) in the form of egg white solid with up to four oral food challenges as directed by protocol.
  Interventions: Drug: Egg Oral Immunotherapy

INTERVENTIONS:
Drug: Egg Oral Immunotherapy — Commercially available egg white solid dispensed by the central manufacturer. Study product will be dispensed in vials for low doses, capsules for mid-range doses, and bulk powder with dosing scoops for the higher doses.
  Other Names: Egg white solid
  Arms: Egg OIT Assigned; Egg OIT Randomized
Drug: Baked Egg — Predetermined food substances with known amounts of Baked Egg (egg protein) with standardized dosing/consumption instructions.
  Arms: Baked Egg Randomized

SUMMARY:
The purpose of this study is to compare Baked Egg vs. Egg Oral Immunotherapy for inducing sustained unresponsiveness to egg exposure in children.

DETAILED DESCRIPTION:
Food allergy affects 6-8 percent of children in the United States. In young children, reactions to egg can range from hives to severe life threatening allergic reactions called anaphylaxis. Current treatment for food allergy is complete avoidance of the food and to carry antihistamines and self-injectable epinephrine if an accidental reaction occurs. However, accidental exposure to allergens in processed foods may be difficult to avoid. Currently, several therapeutic strategies are being investigated to prevent and treat food allergies. Since immunotherapy injections for food allergy are associated with a high rate of allergic reactions, alternate approaches to treatment are needed. Oral (by mouth) immunotherapy (OIT) is one approach that has been tried in some studies in the treatment of food allergies. The purpose of this study is to compare baked foods with egg versus (vs.) egg OIT. The intent of the study is to investigate if participants will be able to consume egg after taking baked foods with egg or egg OIT for a period of time and then stopping for a certain period. This is referred to as tolerance or sustained unresponsiveness. This study will evaluate the effectiveness of the egg OIT vs. baked egg by having each participant ingest egg white solid or baked foods with egg. This will be done over 2 years.

This study will last 2 years. All eligible subjects will receive a baked egg oral food challenge (OFC). Those who pass the baked egg OFC will then have a 2 gm egg OFC. Those who react to the egg OFC will be randomized to Baked Egg or Egg OIT. Individuals who do not pass the initial baked egg OFC will be assigned to Egg OIT. Those who pass the egg OFC will not be eligible for the study and will be followed per site standard of care. All eligible and enrolled subjects will have a 1-year and a 2-year OFC.

At selected visits, blood and urine collection, physical examination, prick skin tests, and atopic dermatitis and asthma evaluations will occur.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 through 16 years with a serum IgE to egg of >= 5 kUA/L within the past 12 months]
* Reacting to the initial baked egg OFC with dose limiting symptoms OR
* Reacting on a 2 gm egg OFC with dose limiting symptoms to a cumulative dose of 2 gm or less after passing the initial baked egg OFC
* Written informed consent from subject and/or parent/guardian
* Written assent from all subjects as appropriate
* All females of child bearing age must be using appropriate birth control

Exclusion Criteria:

* History of anaphylaxis to egg resulting in hypotension, neurological compromise or mechanical ventilation
* Chronic disease (other than asthma, atopic dermatitis, rhinitis) requiring therapy (e.g., heart disease, diabetes)
* Active eosinophilic gastrointestinal disease in the past 2 years
* Participation in any interventional study for the treatment of food allergy in the past 6 months
* Subject is on "build-up phase" of immunotherapy (i.e., has not reached maintenance dosing). Subjects tolerating maintenance allergen immunotherapy can be enrolled.
* Severe asthma, or uncontrolled mild or moderate asthma. More information on these exclusion criteria can be found in the protocol.
* Inability to discontinue antihistamines for initial day escalation, skin testing or OFC
* Use of omalizumab or other non-traditional forms of allergen immunotherapy (e.g., oral or sublingual) or immunomodulator therapy (not including corticosteroids) or biologic therapy (e.g. infliximab, rituximab, etc.) within the past year
* Use of Beta-blockers (oral), angiotensin-converting enzyme (ACE) inhibitors, angiotensin-receptor blockers (ARB) or calcium channel blockers
* Use of investigational drug within 90 days or plan to use investigational drug during the study period
* Pregnancy or lactation

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2013-07; Primary Completion 2017-09-28 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh A Sampson, MD, Study Chair — Icahn School of Medicine at Mount Sinai; Robert Wood, MD, Principal Investigator — Johns Hopkins University
Locations (5):
- United States (5):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - National Jewish Health, Denver, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina

REFERENCES:
- See also: Study Web Site — http://www.cofargroup.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment began in July 2013 and accrual closed in August 2015.
Period: Overall Study
Arm/Group | Baked Egg Randomized | Egg OIT Randomized | Egg OIT Assigned
Started | 28 | 24 | 40
Initiatiated Treatment | 27 | 23 | 39
Year 1 Desensitization OFC (OFC = oral food challenge) | 23 | 20 | 34
Year 2 Desensitization OFC (Completed Year 2 desensitization oral food challenge) | 19 | 20 | 33
Year 2 Sustained Unresponsiveness OFC (Completed Year 2 sustained unresponsiveness oral food challenge (SU OFC)) | 4 | 18 | 21
Completed | 19 | 20 | 32
Not Completed | 9 | 4 | 8
Not completed — Withdrew prior to treatment | 1 | 1 | 1
Not completed — Dosing Symptoms | 1 | 2 | 6
Not completed — Withdrawal by Subject | 5 | 0 | 0
Not completed — Non-compliance | 1 | 1 | 0
Not completed — Developed Eosinophilic Esophagitis (EoE) | 1 | 0 | 0
Not completed — Refused SU OFC | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Only treated participants are included in analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Baked Egg Randomized | Egg OIT Randomized | Egg OIT Assigned | Total
Number analyzed (Participants) | 27 | 23 | 39 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.2 (3.0) | 9.1 (3.1) | 8.8 (2.4) | 8.4 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 14 | 32
  Male | 15 | 17 | 25 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 3
  White | 23 | 18 | 31 | 72
  More than one race | 1 | 1 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic or Non-Latino origin | 25 | 23 | 39 | 87
  Hispanic or Latino origin | 2 | 0 | 0 | 2
Other Food Allergy History [Count of Participants; unit: Participants]
  No/Unknown | 1 | 3 | 8 | 12
  Yes | 26 | 20 | 31 | 77
Asthma Severity History [Count of Participants; unit: Participants]
  No History | 9 | 10 | 13 | 32
  Mild intermittent | 16 | 10 | 24 | 50
  Mild persistent | 1 | 2 | 2 | 5
  Moderate persistent | 1 | 1 | 0 | 2
Allergic GI Disease [Count of Participants; unit: Participants] | 0 | 0 | 0 | 0
Allergic Rhinitis [Count of Participants; unit: Participants] | 24 | 18 | 31 | 73
Atopic Dermatitis History [Count of Participants; unit: Participants] | 18 | 13 | 24 | 55
Atopic Dermatitis Score [Median (Inter-Quartile Range); unit: units on a scale] — The Atopic Dermatitis Total Score is scored on a 10 point scale of 0 to 9 where a higher score indicates increasing severity of atopic dermatitis. This score is a combination of three scores that range from 0 to 3 in the following areas: body surface area score, disease course, and disease intensity.
  units on a scale | 0.0 [0 to 5.0] | 0.0 [0 to 5.0] | 0.0 [0 to 4.0] | 0.0 [0 to 5.0]
Baseline Egg IgE [Median (Inter-Quartile Range); unit: kUA/L] — Assay limits of detection Ranges: 0.01 to 100 kUA/L, Values outside of range were truncated (lower and upper values): 0.05 and 101 kUA/L Population: One participant in Egg OIT Assigned arm had no plasma
  kUA/L
    number analyzed (Participants) | 27 | 23 | 38 | 88
    (all) | 9.77 [6.54 to 27.10] | 12.30 [9.09 to 31.10] | 26.25 [11.7 to 68.80] | 15.60 [8.22 to 37.65]
Baseline Total IgE [Median (Inter-Quartile Range); unit: kUA/L] — Assay limits of detection ranges: Total IgE: 5000 kU/L upper limit, Values above range were truncated: 5001 kU/L Population: One participant in Egg OIT Assigned arm had no plasma
  kUA/L
    number analyzed (Participants) | 27 | 23 | 38 | 88
    (all) | 809.00 [389.00 to 1870.00] | 873.00 [269.00 to 1671.00] | 960.00 [390.00 to 1659.00] | 885.50 [366.50 to 1699.00]
Baseline Egg IgG4 [Median (Inter-Quartile Range); unit: mgA/L] — Assay limits of detection ranges: 0.07 to 30 mgA/L, Values outside of range were truncated (lower and upper values): 0.035 and 31 mgA/L Population: One participant in Egg OIT Assigned arm had no plasma
  mgA/L
    number analyzed (Participants) | 27 | 23 | 38 | 88
    (all) | 0.84 [0.08 to 7.31] | 0.81 [0.26 to 3.71] | 0.28 [0.13 to 1.02] | 0.64 [0.17 to 1.84]
Baseline Egg %IgE [Median (Inter-Quartile Range); unit: % IgE] — Population: One participant in Egg OIT Assigned arm had no plasma
  % IgE
    number analyzed (Participants) | 27 | 23 | 38 | 88
    (all) | 1.86 [0.89 to 3.62] | 1.80 [0.97 to 5.29] | 3.06 [1.21 to 5.86] | 2.13 [1.03 to 4.29]
Baseline Ratio IgG4/IgE [Median (Inter-Quartile Range); unit: ratio] — Population: One participant in Egg OIT Assigned arm had no plasma
  ratio
    number analyzed (Participants) | 27 | 23 | 38 | 88
    (all) | 24.94 [2.23 to 119.64] | 25.75 [11.13 to 86.55] | 5.01 [2.79 to 11.24] | 11.18 [3.86 to 42.25]
Baseline Ovalbumin IgE [Median (Inter-Quartile Range); unit: kUA/L] — Assay limits of detection ranges: 0.01 to 100 kUA/L, Values outside of range were truncated (lower and upper values): 0.05 and 101 kUA/L Population: One participant in Egg OIT Assigned arm had no plasma
  kUA/L
    number analyzed (Participants) | 27 | 23 | 38 | 88
    (all) | 5.53 [3.20 to 20.20] | 5.85 [3.41 to 10.40] | 16.10 [7.30 to 29.70] | 8.88 [4.11 to 20.20]
Baseline Ovomucoid IgE [Median (Inter-Quartile Range); unit: kUA/L] — Assay limits of detection ranges: 0.01 to 100 kUA/L, Values outside of range were truncated (lower and upper values): 0.05 and 101 kUA/L Population: One participant in Egg OIT Assigned arm had no plasma
  kUA/L
    number analyzed (Participants) | 27 | 23 | 38 | 88
    (all) | 6.94 [1.52 to 13.40] | 6.93 [3.27 to 13.20] | 16.40 [6.11 to 35.50] | 9.76 [3.48 to 18.95]
Baseline Ovalbumin IgG4 [Median (Inter-Quartile Range); unit: mgA/L] — Assay limits of detection ranges: 0.07 to 30 mgA/L, Values outside of range were truncated (lower and upper values): 0.035 and 31 mgA/L Population: One participant in Egg OIT Assigned arm had no plasma
  mgA/L
    number analyzed (Participants) | 27 | 23 | 38 | 88
    (all) | 0.64 [0.14 to 5.23] | 0.53 [0.09 to 1.93] | 0.33 [0.16 to 1.04] | 0.49 [0.14 to 1.93]
Baseline Ovomucoid IgG4 [Median (Inter-Quartile Range); unit: mgA/L] — Assay limits of detection ranges: 0.07 to 30 mgA/L, Values outside of range were truncated (lower and upper values): 0.035 and 31 mgA/L Population: One participant in Egg OIT Assigned arm had no plasma
  mgA/L
    number analyzed (Participants) | 27 | 23 | 38 | 88
    (all) | 0.25 [0.04 to 1.34] | 0.15 [0.04 to 2.49] | 0.09 [0.04 to 0.26] | 0.11 [0.04 to 0.60]
Baseline Egg Skin Prick Test (SPT) [Median (Inter-Quartile Range); unit: mms] — Skin prick tests performed using study approved procedures for food and environmental allergens. A skin test probe is pressed through a commercial extract of an allergen into the epidermis.
  mms | 7.50 [5.50 to 13.50] | 11.00 [6.50 to 15.00] | 12.00 [7.50 to 16.50] | 11.00 [6.50 to 15.00]
Baseline Milk SPT [Median (Inter-Quartile Range); unit: mms] | 1.00 [0 to 10.00] | 3.00 [0 to 8.50] | 3.50 [0 to 44.00] | 2.50 [0 to 44.00]
Baseline Peanut SPT [Median (Inter-Quartile Range); unit: mms] — Population: One Egg OIT Assigned subject refused to complete the peanut SPT at baseline
  mms
    number analyzed (Participants) | 27 | 23 | 38 | 88
    (all) | 10.50 [3.50 to 17.00] | 11.00 [8.50 to 17.50] | 10.50 [1.75 to 21.00] | 11.00 [3.25 to 17.50]
Baseline Tree SPT [Median (Inter-Quartile Range); unit: mms] | 2.50 [0 to 7.00] | 4.50 [0 to 8.50] | 3.00 [0 to 6.50] | 3.50 [0 to 7.00]
Baseline Grass SPT [Median (Inter-Quartile Range); unit: mms] | 4.50 [0 to 7.00] | 0.00 [0 to 6.50] | 2.50 [0 to 6.50] | 2.50 [0 to 6.50]
Baseline Weed SPT [Median (Inter-Quartile Range); unit: mms] | 1.50 [0 to 5.50] | 0.00 [0 to 3.50] | 0.00 [0 to 3.50] | 0.00 [0 to 4.00]
Baseline Mold SPT [Median (Inter-Quartile Range); unit: mms] | 0.50 [0 to 4.00] | 1.00 [0 to 4.50] | 0.00 [0 to 3.50] | 0.00 [0 to 3.50]
Baseline Cockroach SPT [Median (Inter-Quartile Range); unit: mms] | 0.00 [0 to 1.50] | 0.00 [0 to 3.00] | 0.00 [0 to 2.50] | 0.00 [0 to 2.50]

OUTCOME MEASURES:

1. Primary Outcome: Sustained Unresponsiveness to Egg Consumption at 2 Years.
Description: Sustained unresponsiveness - able to successfully consume 7444 mg egg white protein in a desensitization OFC and, after an 8-10 week egg-free interval, were also able to successfully consume 7444 mg egg white protein in an OFC after up to 2 years of therapy.
Time Frame: 2 Years
Population: All treated participants were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Baked Egg Randomized | Egg OIT Randomized | Egg OIT Assigned
Number analyzed (Participants) | 27 | 23 | 39
Participants | 3 | 10 | 7
Statistical Analysis 1: Comparison: Baked Egg Randomized vs Egg OIT Randomized; % participants passed Year 2 SU OFC: Baked vs. Egg OIT-Randomized; Test type: Superiority; p = 0.009, Barnard's Exact Test; Risk Difference (RD) = 32.4, 95% CI 2-sided [8.9 to 55.8]
Statistical Analysis 2: Comparison: Egg OIT Randomized vs Egg OIT Assigned; % participants passed Year 2 SU OFC: Egg OIT-Randomized vs. Egg OIT-Assigned; Test type: Superiority; p = 0.031, Barnard's Exact Test; Risk Difference (RD) = 25.5, 95% CI 2-sided [2.0 to 49.1]

2. Secondary Outcome: Desensitization to >= 4.444 Grams Egg White Solid.
Description: Development of desensitization to able to successfully consume >=4444 mg egg white protein during a desensitization OFC on therapy at 1 year and 2 years.
Time Frame: 1 Year and 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Baked Egg Randomized | Egg OIT Randomized | Egg OIT Assigned
Number analyzed (Participants) | 27 | 23 | 39
Participants
  Desensitized Success at Year 1 | 8 | 17 | 22
  Desensitized Success at Year 2 | 6 | 20 | 27
Statistical Analysis 1: Comparison: Baked Egg Randomized vs Egg OIT Randomized; % participants desensitized to >=4444 mg at Year 2 OFC: Baked vs. Egg OIT-Randomized; Test type: Superiority; p < 0.0001, Barnard's Exact Test; Risk Difference (RD) = 64.7, 95% CI 2-sided [43.9 to 85.6]
Statistical Analysis 2: Comparison: Egg OIT Randomized vs Egg OIT Assigned; % participants desensitized to >=4444 mg at Year 2 OFC: Egg OIT-Randomized vs. Egg OIT-Assigned; Test type: Superiority; p = 0.151, Barnard's Exact Test; Risk Difference (RD) = 17.7, 95% CI 2-sided [-2.3 to 37.7]
Statistical Analysis 3: Comparison: Baked Egg Randomized vs Egg OIT Randomized; % participants desensitized to >=4444 mg at Year 1 OFC: Baked vs. Egg OIT-Randomized; Test type: Superiority; p = 0.002, Barnard's Exact Test; Risk Difference (RD) = 44.3, 95% CI 2-sided [19.4 to 69.2]
Statistical Analysis 4: Comparison: Egg OIT Randomized vs Egg OIT Assigned; % participants desensitized to >=4444 mg at Year 1 OFC: Egg OIT-Randomized vs. Egg OIT-Assigned; Test type: Superiority; p = 0.181, Barnard's Exact Test; Risk Difference (RD) = 17.5, 95% CI 2-sided [-6.3 to 41.3]

3. Secondary Outcome: Incidence of All Serious Adverse Events
Description: Incidence of all serious adverse events during the study.
  No statistical analyses were performed since there were no events in 2 of the 3 treatment groups and only 1 event in the third so it would not be meaningful.
Time Frame: up to 3 years
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Baked Egg Randomized | Egg OIT Randomized | Egg OIT Assigned
Number analyzed (Participants) | 27 | 23 | 39
Participants | 0 | 0 | 1

4. Secondary Outcome: Number of Participants With Unrestricted Consumption of Unbaked Egg
Description: Number of participants who reported consumption of concentrated (unbaked) egg in their diet on the long-term follow-up questionnaire 3 years after randomization, indicating unrestricted consumption of unbaked egg. This is a qualitative questionnaire asking participants about egg in their diet, symptoms, and what treatment they received for their allergic reactions.
Time Frame: 3 years after randomization
Population: Participants who completed the long term follow-up questionnaire 3 years after randomization are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Baked Egg Randomized | Egg OIT Randomized | Egg OIT Assigned
Number analyzed (Participants) | 17 | 19 | 30
Participants | 4 | 14 | 12
Statistical Analysis 1: Comparison: Baked Egg Randomized vs Egg OIT Randomized; % participants with unrestricted consumption of unbaked (concentrated) egg 3 years after randomization: Baked vs. Egg OIT-Randomized; Test type: Superiority; p = 0.003, Barnard's Exact Test; Risk Difference (RD) = -50.2, 95% CI 2-sided [-78.4 to -21.9]
Statistical Analysis 2: Comparison: Egg OIT Randomized vs Egg OIT Assigned; % participants with unrestricted consumption of unbaked (concentrated) egg 3 years after randomization: Egg OIT-Randomized vs. Egg OIT-Assigned; Test type: Superiority; p = 0.023, Barnard's Exact Test; Risk Difference (RD) = 33.7, 95% CI 2-sided [7.2 to 60.1]

5. Other Pre Specified Outcome: Changes in Egg-specific Mechanistic Measures and Skin Prick Test Results.
Description: Changes in egg-specific IgE and IgG4, changes in SPT mean wheal diameters, basophil reactivity, Th2 and Treg values.
Time Frame: 2 Years
Population: Data not reported because these are for tertiary objectives that are exploratory.
Arm/Group | Baked Egg Randomized | Egg OIT Randomized | Egg OIT Assigned
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 3 years, through last clinic visit.
Description: * Unsolicited - collected by non-systematic assessment
  + Solicited (dosing symptoms from daily logs) - collected by systematic assessment
Arm/Group | Baked Egg Randomized | Egg OIT Randomized | Egg OIT Assigned
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/23 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/23 | 1/39
Other Adverse Events (participants affected / at risk) | 27/27 | 23/23 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Baked Egg Randomized (N=27) | Egg OIT Randomized (N=23) | Egg OIT Assigned (N=39)
Pneumonia (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baked Egg Randomized (N=27) | Egg OIT Randomized (N=23) | Egg OIT Assigned (N=39)
Ear pain+ (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Eyelid oedema+ (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Ocular hyperaemia+ (Eye disorders) | 0 (0) | 0 (0) | 2 (3)
Abdominal discomfort* (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal discomfort+ (Gastrointestinal disorders) | 13 (41) | 15 (244) | 31 (2030)
Abdominal pain upper* (Gastrointestinal disorders) | 0 (0) | 5 (7) | 2 (3)
Abdominal pain* (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1)
Abdominal pain+ (Gastrointestinal disorders) | 0 (0) | 3 (5) | 10 (37)
Diarrhoea* (Gastrointestinal disorders) | 2 (2) | 5 (6) | 9 (10)
Diarrhoea+ (Gastrointestinal disorders) | 1 (1) | 2 (3) | 7 (15)
Dyspepsia+ (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (22)
Flatulence+ (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (49)
Gastrointestinal disorder* (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Lip swelling+ (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nausea* (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nausea+ (Gastrointestinal disorders) | 0 (0) | 1 (2) | 6 (28)
Oral discomfort+ (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Oral disorder+ (Gastrointestinal disorders) | 19 (269) | 16 (487) | 36 (895)
Tongue pruritus+ (Gastrointestinal disorders) | 0 (0) | 1 (5) | 2 (2)
Vomiting* (Gastrointestinal disorders) | 3 (3) | 5 (10) | 3 (4)
Vomiting+ (Gastrointestinal disorders) | 5 (9) | 8 (20) | 20 (62)
Chest discomfort+ (General disorders) | 0 (0) | 1 (2) | 3 (16)
Influenza like illness* (General disorders) | 0 (0) | 0 (0) | 2 (2)
Malaise+ (General disorders) | 0 (0) | 0 (0) | 3 (13)
Pyrexia* (General disorders) | 7 (7) | 7 (13) | 12 (22)
Allergy to animal* (Immune system disorders) | 1 (1) | 1 (1) | 4 (6)
Hypersensitivity* (Immune system disorders) | 1 (1) | 3 (3) | 1 (1)
Bronchitis* (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Cellulitis* (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Croup infectious* (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Ear infection* (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Febrile infection* (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Gastroenteritis viral* (Infections and infestations) | 3 (4) | 5 (7) | 8 (11)
Gastroenteritis* (Infections and infestations) | 4 (5) | 2 (3) | 5 (6)
Gastrointestinal viral infection* (Infections and infestations) | 5 (8) | 4 (5) | 5 (9)
Influenza* (Infections and infestations) | 2 (2) | 2 (3) | 4 (5)
Lice infestation* (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Localised infection* (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Otitis media* (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Pharyngitis streptococcal* (Infections and infestations) | 4 (4) | 4 (4) | 5 (6)
Sinusitis* (Infections and infestations) | 2 (3) | 1 (2) | 3 (3)
Upper respiratory tract infection* (Infections and infestations) | 11 (21) | 10 (15) | 11 (15)
Viral infection* (Infections and infestations) | 4 (5) | 6 (8) | 5 (7)
Viral upper respiratory tract infection* (Infections and infestations) | 8 (14) | 5 (10) | 8 (11)
Concussion* (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Headache* (Nervous system disorders) | 0 (0) | 5 (8) | 3 (3)
Headache+ (Nervous system disorders) | 0 (0) | 0 (0) | 2 (16)
Asthma* (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 4 (4) | 4 (5)
Cough* (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 9 (16) | 3 (3)
Cough+ (Respiratory, thoracic and mediastinal disorders) | 4 (14) | 8 (9) | 10 (39)
Nasal congestion* (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Nasal congestion+ (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (9) | 9 (390)
Nasal pruritus+ (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Oropharyngeal discomfort+ (Respiratory, thoracic and mediastinal disorders) | 7 (39) | 12 (166) | 24 (394)
Oropharyngeal pain* (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (3) | 3 (3)
Rhinorrhoea* (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Sneezing+ (Respiratory, thoracic and mediastinal disorders) | 4 (20) | 3 (4) | 17 (59)
Throat irritation+ (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (19)
Wheezing* (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Wheezing+ (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 5 (18)
Dermatitis atopic* (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Eczema* (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Eczema+ (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (24) | 0 (0)
Pruritus+ (Skin and subcutaneous tissue disorders) | 6 (30) | 4 (22) | 20 (368)
Rash papular* (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Rash* (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 1 (1)
Rash+ (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (182) | 5 (29)
Urticaria+ (Skin and subcutaneous tissue disorders) | 9 (31) | 11 (107) | 17 (58)
Flushing+ (Vascular disorders) | 3 (16) | 4 (5) | 10 (24)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT01846208/SAP_000.pdf
  • Study Protocol (2016-02-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT01846208/Prot_001.pdf